CLINICAL TRIAL: NCT05255549
Title: ESWT Treatment in Post-stroke Patients With Triceps Sural: a Feasibility RCT
Brief Title: Feasibility of ESWT Treatment in Post-stroke Patients With Triceps Sural Spasticity
Acronym: Waves2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31032021
Record Dates: First submitted 2022-02-05; First posted 2022-02-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2021-11

CONDITIONS: Stroke
Keywords: Stroke; Triceps Sural Spasticity; Extracorporeal Shockwave Therapy
MeSH Terms: conditions — Stroke | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental)
  Interventions: Procedure: ESWT + Stretching
- Group II (Sham Comparator)
  Interventions: Procedure: ESWT and SHAM + Stretching

INTERVENTIONS:
Procedure: ESWT + Stretching — 3 weeks intervention:
  * 3 sessions of ESWT, once a week
  * 6 sessions of passive stretching, twice a week
  Arms: Group I
Procedure: ESWT and SHAM + Stretching — 3 weeks intervention:
  * 1 sessions of ESWT + 2 sessions of Sham, once a week
  * 6 sessions of passive stretching, twice a week
  Arms: Group II

SUMMARY:
The main objective is to evaluate the feasibility of two different rehabilitation protocols that differed from the number of treatment sessions (1 session of ESWT versus 3 weekly sessions of ESWT), in patients with triceps surae spasticity after stroke. In both arms the other ESWT parameters (types of ESWT, intensity, frequency, location) and stretching sessions are the same.

Secondary objectives: to compare functional performances in these two groups of patients receiving the different rehabilitation protocol with ESWT, using the following parameters:

- Six Minutes walking test (6MWT) ; - Time Up & Go (TUG); - Modified Ashworth scale (MAS); - Lower Extremity Functional Scale (LEFS); - passive ankle range of motion (p-ROM), pain (NRS); and presence of ankle clonus. These parameters are assessed during baseline (T0), after 4 weeks (T1) and after 12 weeks (T2).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of legal age
* Time elapsed since the stroke between 6 and 60 months
* Autonomous or supervised walking with or without aids
* Spasticity of the sural triceps> 1 on the MAS scale

Exclusion Criteria:

* Joint stiffness of the lower limbs due to other pathologies (ex orthopedic or rheumatological);
* Conditions that interfere with evaluation or collaboration in rehabilitation treatment (major psychiatric illnesses, clearly detectable cognitive deficits, severe pre-existing disabilities, sensory disturbances, etc.)
* Focal antispasmodic toxin treatments in the previous 3 months or phenolic blocks in the previous 9 months in the treatment region
* Treatments with central antispasmodic drugs with dosage modifications in the last week of starting treatment
* Individual neurorehabilitation treatments in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Feasibility of two kind treatments proposed | T1 after 4 weeks from T0 (Enrollment)
  The intervention is feasible if at least 80% of the enrolled patients complete the entire treatment foreseen in the allocation group

SECONDARY OUTCOMES:
Change in Walking Resistance | T0 Enrollment, T1 after 4 weeks from T0, T2 after 12 weeks from T0
  6 minute walking test
Change in Level of mobility and balance | T0 Enrollment, T1 after 4 weeks from T0, T2 after 12 weeks from T0
  Timed Up & Go Test
Change in spasticity | T0 Enrollment, T1 after 4 weeks from T0, T2 after 12 weeks from T0
  Modified Ashworth Scale (MAS). Score from 0 to 4, higher scores mean a worse outcome
Change in Passive ROM of the ankle in dorsiflexion | T0 Enrollment, T1 after 4 weeks from T0, T2 after 12 weeks from T0
  Passive ankle Range of Motion (p-ROM)
Change in Leg Pain | T0 Enrollment, T1 after 4 weeks from T0, T2 after 12 weeks from T0
  Numeric Pain Rating Scale (NPRS) Score from 0 to 10, higher scores mean a worse outcome
Change in Ability to carry out activities of daily living | T0 Enrollment, T1 after 4 weeks from T0, T2 after 12 weeks from T0
  Lower Extremity Functional Scale (LEFS). Score from 0 to 80, higher scores mean a better outcome.
Change in triceps clones | T0 Enrollment, T1 after 4 weeks from T0, T2 after 12 weeks from T0
  Presence of ankle clonus

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Testoni, Dr, Principal Investigator — Azienda AUSLRE
Locations (1):
- Operational Unit of Physical Medicine and Rehabilitation AUSL - IRCCS Reggio Emilia, Reggio Emilia, Emilia-Romagna, Italy